CLINICAL TRIAL: NCT02842593
Title: Vascular Responses to High vs Low Repetition Resistance Exercise Training in Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: REB 14-333-1
Record Dates: First submitted 2016-07-15; First posted 2016-07-25 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Weight-Lifting Exercise Program

ARMS (2):
- Resistance exercise training (Experimental): Whole-body resistance exercise training 4x/week for 12 weeks. Either 'lower-repetition, heavier-load' or 'higher-repetition, lighter-load' intervention.
  Interventions: Behavioral: Lower-repetition, heavier-load; Behavioral: Higher-repetition, lighter-load
- Non-exercising control (No Intervention): Continue habitual physical activity for 12 weeks.

INTERVENTIONS:
Behavioral: Lower-repetition, heavier-load — 8-12 reps/set at ~80% 1 repetition maximum
  Arms: Resistance exercise training
Behavioral: Higher-repetition, lighter-load — 20-25 reps/set at ~30% 1 repetition maximum
  Arms: Resistance exercise training

SUMMARY:
This study evaluates the effects of two types of resistance exercise training (higher-repetition, lower load vs lower-repetition, higher load vs control) on regional and local measures of arterial stiffness in trained young men.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-30 years old
* Non-obese (Body mass index less than 30 kg/m2)
* Non-smoker
* Healthy based on questionnaire responses
* Resistance trained (Resistance training > 2 times per week for 2 years, minimum 1 lower body exercise session per week)

Exclusion Criteria:

* Allergies to milk proteins (whey or casein)
* Any acute or chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin- or non-insulin dependent diabetes or other metabolic disorders-all ascertained through medical history screening questionnaires
* Arthritic conditions
* Individuals who consume any analgesic or anti-inflammatory drug(s), prescription or non- prescription, chronically will be excluded
* A history of neuromuscular problems
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Carotid-femoral pulse wave velocity | 12 weeks post exercise training
  Assessed using applanation tonometry

SECONDARY OUTCOMES:
Common carotid artery distensibility | 12 weeks post exercise training
  Assessed using vascular ultrasound
Left ventricular mass | 12 weeks post exercise training
  Assessed using standard echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada